CLINICAL TRIAL: NCT02528149
Title: Renal Arteries Dysplastic Aneurysms: Anatomopathological and Genetic Study
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1308016
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Fibromuscular Dysplasia; Renal Artery Stenosis
Keywords: Fibromuscular Dysplasia; dysplastic renal artery aneurysm; renal artery aneurysms; non atheromatous; dysplastic; anatomopathologic; genetic
MeSH Terms: conditions — Fibromuscular Dysplasia; Renal Artery Obstruction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples and adjacent part and aneurysm of renal aneurysms
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with renal aneurysm: Patient with one or more renal artery aneurysm (RAA) operated and with tissue; adjacent part and aneurysm; cryopreserved. Blood sample performed at day 1.
  Interventions: Procedure: tissue of adjacent part and aneurysm of renal aneurysm; Other: blood sample

INTERVENTIONS:
Procedure: tissue of adjacent part and aneurysm of renal aneurysm — the samples are collected during surgery of renal artery aneurysms. Th tissue is cryopreserved in liquid nitrogen before analysis
Other: blood sample

SUMMARY:
Fibromuscular dysplasia (FMD) is localized structural defects in the arterial wall, whose innate or acquired character is still unknown. This segmental non atheromatous injury, leads to stenosis of the arteries of small and medium caliber. Renal arteries are the most commonly affected with 60-75% of total fibrodysplasia. Three histological subtypes have been described: intimal, medial and peri-medial. They are not mutually exclusive and can be observed in the same patient.

This is a rare blood disease, occurring in children and young adults. In this young population with long life expectancy, these aneurysmal lesion are associated with 10% risk of rupture. To date, no data have shown in the literature that FMD is link to genetic causes, or if there is specific histopathologic lesions for non-atherosclerotic renal artery aneurysms.

To answer these questions, Cardiovascular Surgery Unit of the University Hospital of Saint-Etienne, French national reference center for renal artery surgery, in association with the Reference Center for Rare Vascular Disease in Paris, designed the first study for pathological and genetic characteristics of dysplastic renal artery aneurysms in young patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more Renal artery aneurysm (RAA), not eligible for endovascular treatment, have been operated at the Hospital of Saint-Etienne, with tissue (adjacent part and aneurysm) cryopreserved in liquid nitrogen in renal lab and then sent in genetic lab in Georges Pompidou European Hospital (EHGP ).
* Patient (or parent/person having parental authority) Affiliate or entitled to a social security scheme.
* Signature of patient consent (or parents or holder of parental authority)

Exclusion Criteria:

* Patient not included in the tissue collection in Georges Pompidou European Hospital (EHGP ).
* Patient refusing to participate in the study and / or genetic analysis or, for juvenile patients, parents or holder of parental authority refusing the minor patient to be involved in the study and / or genetic analysis.
* Patient with FMD whose samples in the tissue collection did not concern aneurysm.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with one or more Renal artery aneurysm (RAA), not eligible for endovascular treatment, have been operated at the Hospital of Saint-Etienne, with tissue (adjacent part and aneurysm) cryopreserved in liquid nitrogen in renal lab and then sent in genetic lab in EHGP.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
anatomopathological characteristics of renal aneurysms | day 1
  Anatomopathological criteria is a composite outcome : Presence of a media thickness, the media disappearance zones, loss of smooth muscle cells (SMC) in the media with replacement by fibrosis, disorganization of SMC, aneurysms, dissections, discontinuity of the internal elastic lamina, and intimal thickening due to myointimal hyperplasia, abnormalities of proteins of the extracellular matrix.

SECONDARY OUTCOMES:
genetic markers in blood samples | day 1
  identify specific genetic markers (mutation, variant) to characterize genes involved in fibromuscular dysplasia
genetic markers in aneurysm tissue | day 1
  identify specific genetic markers (mutation, variant) to characterize genes involved in fibromuscular dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Barral, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (17):
- France (17):
  - CH Henri Mondor, Aurillac
  - CH Louis Pasteur, Bagnols-sur-Cèze
  - CHU Saint-Jacques, Besançon
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Clinique Saint-Germain, Brive-la-Gaillarde
  - Centre Hospitalier A. Gayraud, Carcassonne
  - CH W. Morey, Chalon-sur-Saône
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CH Emile Roux, Le Puy-en-Velay
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital de la mère et de l'enfant, Limoges
  - Hôpital Robert Schuman, Metz
  - Hôpital Lapeyronie, Montpellier
  - CHU Nantes, Nantes
  - CH Niort, Niort
  - Hôpital Européen Georges Pompidou, Paris
  - CHRU Tours, Tours